CLINICAL TRIAL: NCT00340093
Title: The Diabetes Management Study
Brief Title: Diabetes Management Personal Trainer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999902290; 02-CH-N290
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-03-06

CONDITIONS: Diabetes
Keywords: Adherence; Behavioral Intervention; Adolescence; Self-Regulation; Behavioral Medicine; Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Self-Control

INTERVENTIONS:
Behavioral: Managing Diabetes

SUMMARY:
This 1-year study will test the feasibility and effectiveness of a diabetes personal trainer in helping youth with diabetes manage their treatment. It will examine how families with a diabetic child handle the responsibilities of managing diabetes and deal with the changes that come with managing the illness as the child grows up.

Children between 11 and 16 years of age receiving treatment for diabetes type 1 at Johns Hopkins University Medical Center may be eligible for this study. The children must have been diagnosed with diabetes at least 1 year before entering the study and must require insulin treatment. One parent of each child will also participate.

On entering the study, each child and parent will be interviewed about various topics having to do with taking care of diabetes. After the interview, the children will be randomly assigned to one of two groups: Group 1 will receive education information about diabetes management; Group 2 will be enrolled in a program in which they meet with a diabetes personal trainer 6 to 7 times over 2 months for individualized instruction in planning and evaluating their diabetes care activities. They will also keep in contact with their trainer by telephone.

Children in Group 2 will be given a hand-held personal computer device in which they will keep a record of all diabetes-related activities for 3 days, including insulin shots, meals and snacks. In addition, they will wear an accelerometer, a small device that keeps track of the amount of movement they make. At the end of each of the 3 days, the child will complete a 20- to 30-minute telephone interview reviewing the day. They will have a tape-recorded interview about their experiences in taking care of diabetes. Their meetings with the personal trainer also may be taped.

Children in both groups will continue to see the doctor at the clinic as they normally would.

At 2 and 6 months after starting the study, children in both groups will complete a telephone interview about diabetes management. At 12 months they will complete an in-person interview.

DETAILED DESCRIPTION:
Management of diabetes is a complex process involving the conduct of daily self-care activities, problem-solving, and decision-making. Even in the most supportive environment, adherence to the daily regimen is difficult. Adherence is typically lowest among adolescents, who are taking increasing amounts of responsibility for their diabetes management while still maturing cognitively and socially. This pilot study will investigate the feasibility and effectiveness of a personal diabetes trainer in promoting adherence among early adolescents. A sample of 120 youth ages 11 to 16 will be randomized to informational control or a diabetes personal trainer intervention. Measures of adherence, adjustment, conflict, attitudes, and parental involvement will be obtained at baseline, two months, six months, and one year following. Measures of glycemic control will be abstracted from the medical records.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria include 1) youth diagnosed with Type 1 diabetes for a minimum of 1 year and requiring insulin treatment, 2) youth age 11-16, and 3) both youth and a parent with whom the youth lives most of the time and has primary responsibility for child's health willing to participate.

EXCLUSION CRITERIA:

Exclusion criteria include 1) comorbid chronic illness requiring daily medical management or psychiatric diagnosis or 2) youth or parent non-English speaking/writing.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0
Dates: Start 2002-08-23; Study Completion 2007-03-06

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Mount Washington Pediatric Hospital, Baltimore, Maryland

REFERENCES:
- [Background] Brown SA. Effects of educational interventions in diabetes care: a meta-analysis of findings. Nurs Res. 1988 Jul-Aug;37(4):223-30. PMID 3293025